CLINICAL TRIAL: NCT01287026
Title: Real-Time MRI Right Heart Catheterization Using Passive Catheters
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110091; 11-H-0091
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-03-21

CONDITIONS: Caridovascular Disease; Congenital Heart Disease; Pulmonary Hypertension
Keywords: MRI Catheterization; Right Heart Catheterization; Pulmonary Artery Catheterization; MRI Safety; Jugular Vein Catheterization; Heart Catheterization; Heart Disease; Cardiovascular Disease
MeSH Terms: conditions — Heart Defects, Congenital; Hypertension, Pulmonary; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Open Label
  Interventions: Procedure: Cardiac Real-time MRI RHC (Right Heart Catheterization)

INTERVENTIONS:
Procedure: Cardiac Real-time MRI RHC (Right Heart Catheterization)

SUMMARY:
Background:

- Currently, heart catheterization procedures are guided by X-rays. Researchers are developing new techniques to perform heart catheterization without the use of X-rays by investigating possible uses of magnetic resonance imaging (MRI) scans. To study these uses, researchers are interested in performing a part of the standard X-ray catheterization procedure using MRI on individuals who are scheduled to have heart catheterization.

Objectives:

- To examine the safety and feasibility of right-heart catheterization using MRI-guided catheters.

Eligibility:

- Individuals at least 21 years of age who are undergoing a medically necessary heart catheterization procedure.

Design:

* The research MRI procedure will be performed either before or after standard X-ray guided heart catheterization.
* Participants will be transferred from an X-ray table onto an MRI table and advanced into the scanner. Under MRI guidance, a MRI-compatible catheter will be used to measure blood pressure and blood oxygen levels in the heart, and MRI scanning will be performed for approximately 30 minutes.

DETAILED DESCRIPTION:
Heart catheterization is a minimally invasive procedure to measure pressure and inject dye into specific heart cavities. Heart catheterization usually uses X-ray guidance, which involves radiation exposure and which fails to visualize soft tissue.

We have developed real-time magnetic resonance imaging (MRI) to guide heart catheterization with tissue visualization but without X-ray radiation. In the first phase of this protocol we showed that comprehensive right-sided heart catheterization is feasible in adult patients, using commercially available MRI-compatible ( passive ) catheters.

In the second phase of the protocol, we began performing systematic right-sided heart catheterization without X-ray whenever possible. We will assess the hearts response to hemodynamic provocation during MRI catheterization tailored to the patient s problem. We will use this protocol to further refine the technique

If successful, this will enable future testing of devices for adult and pediatric MRI-guided catheterization, such as special active wire guides, which may lead to new non-surgical treatments of cardiovascular disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 2 years old

Undergoing medically necessary diagnostic or interventional right and/or left cardiovascular catheterization

EXCLUSION CRITERIA :

Cardiovascular instability including ongoing acute myocardial infarction, refractory angina or ischemia, and decompensated congestive heart failure.

Women who are pregnant or nursing

Unable to undergo magnetic resonance imaging:

* Cardiac pacemaker or implantable defibrillator
* Cerebral aneurysm clip
* Neural stimulator (e.g. TENS-Unit)
* Any type of ear implant
* Ocular foreign body (e.g. metal shavings)
* Metal shrapnel or bullet.
* Any implanted device (e.g. insulin pump, drug infusion device), unless it is labeled safe for MRI

EXCLUSION CRITERIA FOR GADOLINIUM-BASED CONTRAST AGENTS FOR ADULTS:

Renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m(2) body surface area according to the Modification of Diet in Renal Disease criteria

Glomerular filtration rate will be estimated using the CKD-EPI equation (33):

eGFR equal 141 x (minimum of (Scr/K, 1)(a) x (maximum of (Scr/K, 1)) (-1.209) x 0.993(Ag x 1.018 (if female) x 1.159 (if black)

Where<TAB>Scr equal serum creatinine

a = -0.329 for females and -0.411 for males

k = 0.7 for females and 0.9 for males

Subjects meeting this exclusion criterion may still be included in the study but may not be exposed to gadolinium-based contrast agents.

EXCLUSION CRITERIA FOR GADOLINIUM-BASED CONTRAST AGENTS FOR CHILDREN

Renal excretory dysfunction, estimated glomerular filtration rate < 30 mL/min/1.73m(2) body surface area according to the Schwartz equation for estimation of GFR in children as recommended by the National Kidney Disease Education Program. The Schwartz equation is commonly used for GFR determination in children at Children s National Medical Center, Washington, DC.

GFR (mL/min/1.73 m2) = (k (SqrRoot) height) / serum creatinine concentration where K = constant defined as

follows:

k = 0.33 in premature infants [Excluded from this protocol]

k = 0.45 in term infants to 1 year of age [Excluded from this protocol]

k = 0.55 in children to 13 years of age

k = 0.70 in adolescent males (not females because of the presumed increase in male muscle mass,

the constant remains 0.55 for females)

* Height in cm
* Serum creatinine in mg/dL

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02-23; Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
To test the initial safety and feasibility of diagnostic right heart catheterization in human subjects using MRI- guidance and | Ongoing
  There will be no heating or adverse events related to the MRI RHC.

SECONDARY OUTCOMES:
To train staff in the conduct of simple MRI catheterization in humans, to accrue incremental experience towards more complex MRI catheterization procedures | Ongoing
To test incremental MRI scanning techniques (technical developments) to assist MRI catheterization in humans | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Rogers T, Ratnayaka K, Khan JM, Stine A, Schenke WH, Grant LP, Mazal JR, Grant EK, Campbell-Washburn A, Hansen MS, Ramasawmy R, Herzka DA, Xue H, Kellman P, Faranesh AZ, Lederman RJ. CMR fluoroscopy right heart catheterization for cardiac output and pulmonary vascular resistance: results in 102 patients. J Cardiovasc Magn Reson. 2017 Jul 27;19(1):54. doi: 10.1186/s12968-017-0366-2. PMID 28750642